CLINICAL TRIAL: NCT01531127
Title: Executive Function in Learning in Children With Attention Deficit Hyperactivity Disorder (ADHD) Receiving Medical Treatment Alone Compared to Children Receiving Additional Treatment to Improve Learning Strategies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0014-12-HYMC
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Combined Therapy: ADHD Medication and Learning Strategies Treatment
- ADHD Medication Treatment: Control group

SUMMARY:
The purpose of this study is to determine whether there is a difference in executive function in learning in children with ADHD receiving medical treatment alone to the executive function in children receiving, in addition to medical treatment in learning strategies.

ELIGIBILITY:
Inclusion Criteria:

* Normal development for age
* ADHD

Exclusion Criteria:

* Low compliance
* Developmental delay
* Chronic disease

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ADHD treated in the Institute for Child Development at Hillel Yaffe Medical Center
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Level of Executive Functioning | One year
  Brief Behavior Rating Inventory of Executive Function will be administered

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel